CLINICAL TRIAL: NCT01554215
Title: Phase 1 of Mom Power: Attachment Based Parenting and Self-Care Skills Program
Brief Title: Mom Power is an Attachment Based Parenting Program for Families and Their Children
Acronym: MP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Maria Muzik, Perinatal Psychiatrist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mom Power
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2012-03

CONDITIONS: Parenting
Keywords: parenting; child behavior; attachment
MeSH Terms: conditions — Child Behavior | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mom Power Intervention Group (Experimental): Participants that are randomly assigned to be in the intervention group will be invited to learn about parenting and self-care skills information at a community location, facilitated by two trained and experienced clinicians in a group setting. They will benefit from the en-vivo experience of being supported as a parent and will receive feedback and support about their challenges and strengths in parenting.
  Interventions: Behavioral: Mom Power Intervention Group
- Mom Power Attentional Control Group (Active Comparator): Participants randomly assigned to this group will receive parenting and self-care skills information through the mail weekly.
  Interventions: Behavioral: Mom Power Attentional Control Group

INTERVENTIONS:
Behavioral: Mom Power Intervention Group — attachment-based parenting program for parents in community setting led by trained and experienced facilitators.
  Other Names: attachment; mom power; intervention group
  Arms: Mom Power Intervention Group
Behavioral: Mom Power Attentional Control Group — at home control, weekly mailings
  Other Names: attachment; attentional control; at home control; parenting
  Arms: Mom Power Attentional Control Group

SUMMARY:
Mom Power is a weekly attachment based parenting program aimed to increase parenting and self-care skills for families.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages 15+ years with at least one child , interested in learning about parenting and willing to attend weekly sessions in group setting.
* Participants must be willing to be both videotaped and audio taped for research purposes
* must speak English as their first language.

Exclusion Criteria:

* Participants with no children 0-6 or younger than 15. Participants not willing to attend weekly sessions or participate in group/at home control.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Psychopathology | 3 months
  participants are asked to complete questionnaires related to psychopathology such as depression, anxiety, and post traumatic stress.

SECONDARY OUTCOMES:
Parenting | 3 months
  Measures looking at parental bonding, parenting self-efficacy and feelings of helplessness will be assessed. In addition, videotaped sessions of parent and child engaging in play will be coded and assessed.
Maternal Mental Representations | 3 months
  Participants participate in a structured interview asking about their relationship with their child. Interviews are coded and classified relating to attachment style.
Connection to Care | 3 months
  Participants will be referred to community agencies for resources based on need during their involvement with Mom Power. The referrals, follow-up with referrals and health care utilization will be tracked to determine engagement with resources.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Muzik, MD, Principal Investigator — University of Michigan Department of Psychiatry
Locations (1):
- University of Michigan Department of Psychiatry, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Jester JM, Riggs JL, Menke RA, Alfafara E, Issa M, Muzik M, Rosenblum KL. Randomized pilot trial of the "Mom Power" trauma- and attachment-informed multi-family group intervention in treating and preventing postpartum symptoms of depression among a health disparity sample. Front Psychiatry. 2023 Sep 5;14:1048511. doi: 10.3389/fpsyt.2023.1048511. eCollection 2023. PMID 37732075
- [Derived] Rosenblum KL, Muzik M, Morelen DM, Alfafara EA, Miller NM, Waddell RM, Schuster MM, Ribaudo J. A community-based randomized controlled trial of Mom Power parenting intervention for mothers with interpersonal trauma histories and their young children. Arch Womens Ment Health. 2017 Oct;20(5):673-686. doi: 10.1007/s00737-017-0734-9. Epub 2017 Jun 25. PMID 28647759